CLINICAL TRIAL: NCT00769028
Title: A Double-Blind Placebo-Controlled Pilot Study of Safety and Tolerability of AIMSPRO in Established Diffuse Cutaneous Systemic Sclerosis
Brief Title: AIMSPRO in Established Diffuse Cutaneous Systemic Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daval International Limited (Industry)
Responsible Party: Prof. Christopher Denton, Royal Free Hospital NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DISS01
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Diffuse cutaneous systemic sclerosis; Scleroderma; Biological; Hyperimmune caprine serum; Goat Serum
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AIMSPRO (Experimental)
  Interventions: Drug: Hyperimmune caprine serum
- Placebo (Placebo Comparator)
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: Hyperimmune caprine serum — Subcutaneous injection of serum, 1ml twice weekly for 6 months
  Other Names: Ceremben; Hyperimmune goat serum
  Arms: AIMSPRO
Drug: Albumin — Subcutaneous injection of albumin, 1ml twice weekly for 6 months
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To study the safety and tolerability of a hyperimmune goat serum product (AIMSPRO) in the treatment of systemic sclerosis (SSc) through a period of 26 weeks of study participation. The secondary objective of the study is to assess the efficacy of AIMSPRO as a therapeutic agent for SSc using inter alia the SSc-HAQ questionnaire and the modified Rodnan skin score.

DETAILED DESCRIPTION:
Systemic sclerosis (scleroderma, SSc) is a multisystemic disease clinically characterized by fibrosis of the skin, joints, muscles and internal organs. Systemic sclerosis is a rare disease, with an estimated incidence of 19 individuals per million population per year.

The pathogenesis of SSc remains incompletely understood although it seems likely that there is an interplay between inflammatory, vascular and fibroblast dysfunction, leading ultimately to the sustained activation of a population of fibroblasts that deposit increased amounts of extracellular matrix in lesional tissues, including the skin and internal organs.

Impairment of the immune system is currently thought to play an important role. This is based on the observation that in the early phases of SSc, mononuclear cells migrate to the dermis and accumulate around small blood vessels, nerves and skin appendages. Furthermore, there is a direct relation between the extent of cutaneous inflammation and the extent and progression of fibrosis of the skin. Stimulated T-lymphocytes of patients with SSc produce more tumor necrosis factor-α, interleukin-1 and -2 compared with healthy controls and the serum concentrations of IL-2, IL-4, IL-6 and IL-8 and soluble IL-2 receptors are elevated. The occurrence of autoantibodies, predominantly antitopoisomerase-1 (ATA) and anticentromere antibodies (ACA), in approximately 90% of the patients, points to an alteration of the humoral immune system.

Systemic sclerosis can be subdivided into diffuse and limited forms. Diffuse cutaneous SSc (dcSSc) is characterised by skin involvement proximal to the elbows and knees, limited cutaneous SSc (lcSSc) by skin involvement distal to these joints. In approximately 50% of patients with dcSSc, ATA can be detected, and in approximately 50% of patients with lcSSc ACAs are present. Other hallmark autoantibodies have also been identified in smaller proportions of SSc patients including anti-RNA polymerase I/III and anti-fibrillarin antibodies (5).

The course of SSc is variable. In some patients the disease remains confined to sclerodactyly and Raynaud's phenomenon. In other patients there is a relentless progression of internal organ fibrosis, ultimately leading to death. A recent study showed a cumulative 5-year survival rate of 63%. There are efforts to try to identify clinical and investigational predictors of outcome in SSc. One study has identified three clinical variables: raised ESR, proteinuria and impaired lung function indices which are associated with poor outcome. In addition, the various hallmark autoantibodies occurring in SSc are mutually exclusive and several studies in Europe and North America have demonstrated that individuals carrying each of these autoantibodies are associated with different frequencies of internal organ complications. This also allows patients who are at increased risk of pulmonary, cardiac or renal complications to be identified.

At present, no treatment has been definitely shown to be effective in SSc. Because of its presumed immunologic pathogenesis, modulation of the immune system has been the major goal in therapeutic interventions in SSc. Several studies have reported effectiveness of immune modulating drugs in the treatment of this disease, although these have mostly been in open, uncontrolled trials. These drugs include azathioprine, cyclosporin, methotrexate and cyclophosphamide. Amongst these, methotrexate and cyclophosphamide are currently the most widely used. New, more specific immunological treatment modalities have been harnessed in order to improve the treatment and prognosis of scleroderma patients.

In 2005, a patient with systemic sclerosis was treated with AIMSPRO on a compassionate basis with a sustained improvement in mobility and, in particular, there was an improvement in proximal muscle power and skin characteristics.

In this study, twenty patients will receive either AIMSPRO or placebo, 1.0ml subcutaneously, twice weekly for 26 weeks. Standard outcome measures and novel biomarkers will be used to investigate safety, efficacy and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must fulfill 1980 Preliminary Classification Criteria for systemic sclerosis of the American Rheumatism Association
* Diffuse cutaneous SSc, as evidenced by skin sclerosis proximal to the elbows or knees and absence of the anti-centromere autoantibody
* At least three years must have elapsed since the first non-Raynaud's manifestation
* Men and women of childbearing potential must use adequate birth control measures for the duration of the study and should continue such precautions for six months after receiving the last injection of AIMSPRO.
* Screening laboratory test results:

Hemoglobin > 8.5 g/dL WBC > 3.5 x 10^9/L Neutrophils > 1.5 x 10^9/L Platelets > 100 x 10^9/L SGOT (AST) and alkaline phosphatase levels must be within twice the upper limit of normal range for the laboratory conducting the test.

* Patient must be able to adhere to the study visit schedule and other protocol requirements
* Patient must be capable of giving informed consent and the consent must be obtained prior to any screening procedures
* No radiological evidence of malignancy, infection or (previous) tuberculosis in a chest radiograph performed within three months prior to the first injection of study drug

Exclusion Criteria:

* Women who are pregnant, nursing, or planning pregnancy within one and a half years after screening (i.e., approximately six months following last injection of study drug).
* Use of any investigational drug within one month prior to screening or within five half-lives of the investigational agent, whichever is longer.
* Use of a putative disease modifying drug (potential immunosuppressive drug) within one month of screening.
* Treatment with any therapeutic agent targeted at reducing TNF (e.g., infliximab, pentoxifylline, thalidomide, etanercept, etc.) within three months of screening.
* Previous administration of AIMSPRO.
* History of known allergy to animal proteins.
* Serious infections (such as pneumonia or pyelonephritis) in the previous three months. Less serious infections (such as acute upper respiratory tract infection [colds] or simple urinary tract infection) should be monitored to their conclusion or treated, as appropriate, prior to inclusion.
* Active hepatitis-B or hepatitis-C.
* Active tuberculosis.
* Patients with opportunistic infections, including but not limited to evidence of active cytomegalovirus, active Pneumocystis carinii, Aspergillosis, histoplasmosis or atypical mycobacterium infection, etc, within the previous six months.
* History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infra-clavicular, epitrochlear, or periaortic areas), or splenomegaly.
* Known recent substance abuse (drug or alcohol).
* Poor tolerability of venepuncture or lack of adequate venous access for required blood sampling during the study period.
* Presence of a transplanted organ (with the exception of a corneal transplant > three months prior to screening).
* Patients receiving immunosuppressive therapy within one month of screening.
* Patients with malignancy within the past five years.
* Signs or symptoms of severe, progressive or uncontrolled renal, hepatic, haematologic, gastrointestinal, endocrine, pulmonary, cardiac or neurological disease (including demyelinating diseases such as multiple sclerosis).
* Patients who, within the past three months, have had either a myocardial infarction, uncontrolled congestive cardiac failure, unstable angina, uncontrolled systemic hypotension or uncontrolled systemic hypertension.
* Patients who have screening laboratory values which deviate 20% or more from the upper or lower limits of normal or which are considered to be clinically significant to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Modified Rodnan Skin Score | Baseline, Week 6 and Week 26

SECONDARY OUTCOMES:
Scleroderma Health Assessment Questionnaire | Baseline, Week 6 and Week 26
Scleroderma UK Functional Score | Baseline, Week 6 and Week 26
Patient and Physician Global Assessment (VAS) | Baseline, Week 6 and Week 26
SF-36 (Short form 36) | Baseline, Week 6 and Week 26
MRC Sum Score | Week 0, Week 6 and Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Denton, PhD FRCP, Principal Investigator — Royal Free Hospital NHS Trust
Locations (1):
- Centre for Rheumatology and Connective Tissue Diseases, Lower Ground Floor, Royal Free Hospital NHS Trust, Hampstead, London, United Kingdom

REFERENCES:
- [Derived] Quillinan N, Clark KE, Youl B, Vernes J, McIntosh D, Haq S, Denton CP. Multiplex serum protein analysis reveals potential mechanisms and markers of response to hyperimmune caprine serum in systemic sclerosis. Arthritis Res Ther. 2017 Mar 7;19(1):45. doi: 10.1186/s13075-017-1252-x. PMID 28270187
- [Derived] Quillinan NP, McIntosh D, Vernes J, Haq S, Denton CP. Treatment of diffuse systemic sclerosis with hyperimmune caprine serum (AIMSPRO): a phase II double-blind placebo-controlled trial. Ann Rheum Dis. 2014 Jan;73(1):56-61. doi: 10.1136/annrheumdis-2013-203674. Epub 2013 Sep 25. PMID 24067785